CLINICAL TRIAL: NCT05444049
Title: A Feasibility Study of the NEURESCUE Device as an Adjunct to In-Hospital Cardiac Arrest
Brief Title: NEURESCUE Device as an Adjunct to In-Hospital Cardiac Arrest (ARISE)
Acronym: ARISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: neurescue (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Safestudy3
Record Dates: First submitted 2022-06-28; First posted 2022-07-05 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2024-10

CONDITIONS: Cardiac Arrest; Cardiopulmonary Arrest; Cardiovascular Diseases
MeSH Terms: conditions — Heart Arrest; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): The NEURESCUE device will be used as an adjunct to ACLS.
  Interventions: Device: NEURESCUE device

INTERVENTIONS:
Device: NEURESCUE device — The balloon catheter is delivered via the femoral artery, temporarily inflating a soft balloon in the descending aorta to redirect blood flow towards the upper body.

SUMMARY:
The NEURESCUE device is the first intelligent catheter for aortic balloon occlusion, an emergency technique that supercharges blood flow to the heart and brain within one minute from deployment.

The catheter-based device is delivered via the femoral artery, temporarily inflating a soft balloon in the descending aorta to redirect blood flow towards the upper body.

The objective of this study is to investigate the feasibility of the NEURESCUE device as an adjunct to Advanced Cardiac Life Support (ACLS) in adults with cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤80 years
2. CPR initiated within 7 min of presumed arrest
3. 8 min of continuous ACLS without ROSC

Exclusion Criteria:

1. Traumatic cardiac arrest
2. Intraoperative cardiac arrest
3. Known pregnancy
4. Known terminal disease
5. Known do-not-attempt-CPR order
6. Subjects whose femoral arterial access site cannot accommodate an 8 Fr introducer sheath
7. Subjects currently on mechanical circulatory support

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Successful balloon inflation within 10 minutes from first vessel puncture | Assessed up to 10 min

SECONDARY OUTCOMES:
Change in central blood pressure | Assessed up to 1 hour
Total ACLS time at initiation of the investigational procedure | Assessed up to 1 hour
Time from first vessel puncture to successful sheath insertion | Assessed up to 1 hour
Rate of occlusion success | Assessed up to 1 hour
Return of spontaneous circulation (ROSC) | Assessed up to 1 hour
  The endpoint is dichotomous (yes/no) for each subject

CONTACTS AND LOCATIONS:
Overall Officials: David Shavelle, M.D., Principal Investigator — Long Beach Medical Center
Locations (1):
- Long Beach Medical Center, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual request